CLINICAL TRIAL: NCT00486746
Title: Lifestyle Intervention Treatment for Patients With Mild Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other); Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Juha Seppa, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5551811
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; lifestyle intervention; cardiovascular
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Exercise; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention (Experimental)
  Interventions: Behavioral: Lifestyle intervention (physical activity and dietary counseling)
- General health counseling (Active Comparator)
  Interventions: Behavioral: General information on healthy lifestyle habits

INTERVENTIONS:
Behavioral: Lifestyle intervention (physical activity and dietary counseling) — One-year intervention
  Arms: Lifestyle intervention
Behavioral: General information on healthy lifestyle habits — A single session
  Arms: General health counseling

SUMMARY:
The main objective of the study is to determine whether a supervised lifestyle intervention including individualized dietary counseling could be a curative treatment for patients with mild OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is one of the most common sleep disturbances, and it has been estimated that one out of five adults has at least some degree of sleep related breathing disturbances. Obstructive sleep apnea affects mostly the middle-aged work force, and causes a negative impact on public health by increasing both morbidity and mortality. Obesity is related to many diseases including diabetes, cardiovascular diseases, and metabolic syndrome,and obesity is also considered as the most important risk factor for OSA.Considering the prevalence of mild OSA, and the beneficial effects of even a slight weight loss on both the severity of OSA and the likelihood of developing OSA, lifestyle intervention including weight reduction represents a viable option for the treatment of patients with mild OSA.However, although included in the clinical guidelines, there is a definite lack of well executed studies on the effect of weight reduction upon OSA. Accordingly, we are conducting a randomized study on the effects of lifestyle intervention in the most prevalent subgroup of OSA patients, overweight patients with mild OSA. The study is an on-going prospective, randomized, parallel group trial. The main objective of the study is to determine whether a supervised lifestyle intervention including individualized dietary counseling could be a curative treatment for patients with mild OSA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Apnea-hypopnea index 5-15
* BMI 28-40

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate, if weight reduction and lifestyle intervention improve the symptoms of mild obstructive sleep apnoea | 3 months
To evaluate, if these favourable changes remain in follow-up. | 1, 2 and 5 years

SECONDARY OUTCOMES:
To evaluate, whether the treatment of mild OSA prevents the development of diseases in general associated with sleep apnoea | 5 years
To evaluate, whether the mild OSA has detrimental effects on cardiovascular functions and glucose-, insulin- and lipid metabolisms, regulation of autonomous nervous system, endothelial function, baroreflex sensitivity | baseline, 3 months, 1, 2 and 5 years
To evaluate, if improvement of mild OSA has beneficial influence on quality of life, cardiovascular functions and glucose-, insulin- and lipid metabolisms, regulation of autonomous nervous system, endothelial function, and anatomy of the pharynx | 1,2,5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henri Tuomilehto, PhD, Study Director — Kuopion University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

REFERENCES:
- [Derived] Tuomilehto H, Seppa J, Uusitupa M, Tuomilehto J, Gylling H; Kuopio Sleep Apnea Group. Weight reduction and increased physical activity to prevent the progression of obstructive sleep apnea: A 4-year observational postintervention follow-up of a randomized clinical trial. [corrected]. JAMA Intern Med. 2013 May 27;173(10):929-30. doi: 10.1001/jamainternmed.2013.389. No abstract available. PMID 23589169
- [Derived] Lehto SM, Sahlman J, Soini EJ, Gylling H, Vanninen E, Seppa J, Viinamaki H, Tuomilehto H. The association between anxiety and the degree of illness in mild obstructive sleep apnoea. Clin Respir J. 2013 Apr;7(2):197-203. doi: 10.1111/j.1752-699X.2012.00304.x. PMID 22686135
- [Derived] Sahlman J, Seppa J, Herder C, Peltonen M, Peuhkurinen K, Gylling H, Vanninen E, Tukiainen H, Punnonen K, Partinen M, Uusitupa M, Tuomilehto H. Effect of weight loss on inflammation in patients with mild obstructive sleep apnea. Nutr Metab Cardiovasc Dis. 2012 Jul;22(7):583-90. doi: 10.1016/j.numecd.2010.10.007. Epub 2010 Dec 28. PMID 21193295
- [Derived] Tuomilehto H, Gylling H, Peltonen M, Martikainen T, Sahlman J, Kokkarinen J, Randell J, Tukiainen H, Vanninen E, Partinen M, Tuomilehto J, Uusitupa M, Seppa J; Kuopio Sleep Apnea Group. Sustained improvement in mild obstructive sleep apnea after a diet- and physical activity-based lifestyle intervention: postinterventional follow-up. Am J Clin Nutr. 2010 Oct;92(4):688-96. doi: 10.3945/ajcn.2010.29485. Epub 2010 Aug 11. PMID 20702607
- [Derived] Kemppainen T, Ruoppi P, Seppa J, Sahlman J, Peltonen M, Tukiainen H, Gylling H, Vanninen E, Tuomilehto H. Effect of weight reduction on rhinometric measurements in overweight patients with obstructive sleep apnea. Am J Rhinol. 2008 Jul-Aug;22(4):410-5. doi: 10.2500/ajr.2008.22.3203. PMID 18702908